CLINICAL TRIAL: NCT01059838
Title: Speech Perception in Noise for Children With Cochlear Implants
Brief Title: Speech Perception for Children With Cochlear Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Cynthia Hogan, PhD, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-005368
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Hearing Loss
Keywords: pediatrics; cochlear implant
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single subject (Experimental)
  Interventions: Behavioral: sentence recognition

INTERVENTIONS:
Behavioral: sentence recognition — testing the ability for sentence recognition in quiet and in noise.

SUMMARY:
The purpose of this study is to determine whether speech recognition in noise can be improved by the addition of a special listening program to the sound processor. Thus we propose to assess speech perception in noise for pediatric cochlear implant patients using both their everyday listening program as well an ASC program.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether speech recognition in noise can be improved by the addition of a special listening program to the sound processor. Thus we propose to assess speech perception in noise for pediatric cochlear implant patients using both their everyday listening program as well an ASC program.

You will be asked to listen to sentences in quiet and in noise and repeat the sentences. You will be seated in a comfortable chair inside the sound booth with 8 loudspeakers placed in a circular pattern around your head. We will test your sentence recognition abilities in your listening program as well as in the new listening program. The sentences and noise will be presented through loudspeakers at levels typically encountered in everyday communication environments. Your participation would involve approximately 20 minutes of testing plus 10 minutes to add the new listening program to their processor.

ELIGIBILITY:
Inclusion Criteria: Children with bilateral sensorineural hearing loss who have 1) one or two Nucleus 24 series cochlear implants, 2) at least 1 year experience with their cochlear implant, and, 3) the ability to score > 50% correct for HINT sentences in quiet.

Exclusion Criteria: 1) Patients under 4 years of age or over 17 years of age, 2) patients who have had at least 1 year experience with their cochlear implant and, 3) patients who score > 50% for HINT sentence recognition in quiet

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The Objective is to examine speech perception performance in the presence of restaurant noise for pediatric cochlear implant recipients in two listening conditions: ADRO alone & ASC + ADRO. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Hargenrader, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States